CLINICAL TRIAL: NCT00123097
Title: Multicenter Trial of CPE for Maxillofacial Prosthetics
Brief Title: Clinical Trial of New Elastomer for Maxillofacial Prosthetics
Status: Completed | Phase: Phase 3 | Type: Interventional
Sponsor: University of Louisville (Other)
Collaborators: National Institute of Dental and Craniofacial Research (NIDCR) (NIH)
Responsible Party: Principal Investigator, Lawrence M. Gettleman, DMD, MSD, Professor, Gratis, University of Louisville
Allocation: Randomized | Model: Crossover | Masking: Quadruple | Purpose: Device Feasibility
Other Study IDs: NIDCR-14543; U01DE014543 (NIH); 5U01DE014543 (NIH); NCT00408486 (obsolete NCT alias)
Record Dates: First submitted 2005-07-21; First posted 2005-07-22 (Estimated); Last update posted 2017-04-07 (Actual); Status verified 2017-04

CONDITIONS: Facial Neoplasms; Head and Neck Neoplasms; Head Injuries, Penetrating; Birth Injuries
Keywords: Facial Neoplasms; Head and Neck Neoplasms; Head Injuries, Penetrating; Birth Injuries
MeSH Terms: conditions — Facial Neoplasms; Head and Neck Neoplasms; Head Injuries, Penetrating; Birth Injuries

STUDY DESIGN:
Who Masked: Participant, Care Provider, Investigator, Outcomes Assessor

ARMS (2):
- Chlorinated polyethylene elastomer first (Experimental): Patient receives prosthetic made from CPE then the SOC, silicon.
  Interventions: Combination Product: Chlorinated polyethylene elastomer
- Silicon first (Active Comparator): Patient receives prosthetic made from the SOC, silicon, followed by the CPE,Chlorinated polyethylene elastomer.
  Interventions: Combination Product: Chlorinated polyethylene elastomer

INTERVENTIONS:
Combination Product: Chlorinated polyethylene elastomer — Chlorinated polyethylene
  Other Names: CPE

SUMMARY:
The purpose of this study is to evaluate a new rubber material used to make prosthetic replacements of the face lost to cancer, trauma, or birth defects.

DETAILED DESCRIPTION:
Maxillofacial prosthetics is a subspecialty of prosthodontics, providing the clinical rehabilitation treatment of patients who have lost parts of the face due to cancer, trauma, or birth defects. It is an orphan field that:

* treats few patients, making the subspecialty unprofitable for manufacturers to develop new materials;
* offers fundamental rehabilitation and improvement in the quality of life to patients who may have exhausted personal or third party funding; and
* provides a dental solution to an essentially medical problem.

Silicone rubber materials have been used for facial rehabilitation for more than 4 decades with few improvements. There is a clear need for new, alternative, and more economic materials for extraoral maxillofacial prostheses. Research at Gulf South Research Institute in New Orleans by the Principal Investigator and others in the 1970s and 1980s developed an alternative low-cost thermoplastic industrial rubber material (chlorinated polyethylene, CPE) that met all toxicological (safety) and physical (effectiveness) requirements. A Phase 2 clinical trial at the time yielded equivocal results when compared to conventional but costly silicone rubber products.

This research is a controlled, randomized, single-crossover, double-blinded investigator-initiated multicenter Phase 3 clinical trial treating 100 patients that evaluates:

* experimental thermoplastic CPE; and
* control silicone (Silastic Adhesive A/MDX4-4210) materials for non-inferiority of CPE based on functional and subjective characteristics, and on the quality of life.

The clinical centers of the trial are at M.D. Anderson Cancer Center in Houston, Texas, and at the Toronto Sunnybrook Regional Cancer Centre in Toronto, Canada.

ELIGIBILITY:
Inclusion Criteria:

* Requires treatment for developmental or acquired extraoral facial defect
* Fully healed wound (6 months after surgery and/or radiation)
* Defect no larger than 9 x 12 cm (3.5 x 4.5 inches, the diameter of a giant bronze flask)
* Cognizant enough to answer questionnaires
* Agrees to wear the prosthesis at least 6 hours per day
* Agrees to use the prescribed adhesive (Epithane-3 - now called Daro Adhesive Extra Strength) and clean and store as instructed
* Plans to be able to return to the research institution for a 10 month period
* Able to manage prosthesis him/herself or with caregiver for a 10 month period
* Karnofsky score greater than or equal to 60 (www.hospicepatients.org/karnofsky.html)
* No framework or implant/magnet retention
* No multiple recurrences of tumor
* No hypersensitivity to adhesives or test materials
* No current systemic or topical facial steroid treatment
* Not legally blind
* Not expected to have further surgeries to defect, radiation therapy, or other cytoreductive therapy over the next 10 months
* No evidence of active skin condition/disease
* Not an infectious risk patient

Min Age: 21 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Enrollment: 42 (Actual)
Dates: Start 2005-02; Primary Completion 2009-08 (Actual); Study Completion 2009-08 (Actual)

PRIMARY OUTCOMES:
Non-inferiority of chlorinated polyethylene elastomer (CPE) material | 10 month

CONTACTS AND LOCATIONS:
Overall Officials: Sudarat Kiat-amnuay, DDS MS, Study Chair — University of Texas Dental Branch; Mark S Chambers, DMD MS, Study Chair — MD Anderson Cancer Center, Dept. of Head & Neck Surgery; James D Anderson, DDS MScD, Principal Investigator — Toronto Sunnybrook Regional Cancer Centre; Lawrence Gettleman, DMD, MSD, Principal Investigator — University of Louisville, School of Dentistry
Locations (1):
- University of Louisville, Louisville, Kentucky, United States

REFERENCES:
- [Derived] Kiat-amnuay S, Jacob RF, Chambers MS, Anderson JD, Sheppard RA, Johnston DA, Haugh GS, Gettleman L. Clinical trial of chlorinated polyethylene for facial prosthetics. Int J Prosthodont. 2010 May-Jun;23(3):263-70. PMID 20552094